CLINICAL TRIAL: NCT06326775
Title: Research on Precision Pharmaceutical Care for Heart Transplant Recipients
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Changhai Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, JunRong zhu, Deputy Director of Pharmacy Department, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20240311-KS-02
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Heart Transplant Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishing personalized dose prediction and related adverse drug reaction prediction models for immunosuppressive drugs after heart transplantation using multiple methods to construct a precise pharmaceutical service system for heart transplant patients has important research value and clinical significance in improving the safety and effectiveness of medication for patients.

DETAILED DESCRIPTION:
In recent years, model-guided precision medication has become synonymous with modern individualized drug therapy methods. Heart transplantation (HT) is the preferred treatment for patients with end-stage heart failure, as it not only improves the quality of life but also extends the patient's lifespan. However, the host's immune response to the allograft after transplantation has always been one of the main factors affecting the short-term and long-term survival rates after heart transplantation. Recipients need to take immunosuppressants for a long time to improve the long-term survival rate of the graft and the recipient. However, there is a significant individual difference in the clinical application of these drugs. Establishing a risk prediction assessment model for drug administration and an evaluation system for pharmacodynamics and adverse events is an urgent clinical issue to be resolved. For example, tacrolimus (TAC) is a macrolide calcineurin inhibitor with strong immunosuppressive properties. More than 93% of heart transplant recipients use TAC to prevent transplant rejection, which is the cornerstone of the triple immunosuppressive regimen. Studies have shown that acute rejection, infection, acute kidney injury, and other complications usually occur in the early stage after heart transplantation and are significantly related to TAC blood concentration levels. Therefore, accurately estimating the individualized dosage of immunosuppressants after transplantation and accurately predicting the risk of various adverse events such as rejection, infection, and acute kidney injury in heart transplant patients after taking immunosuppressants, constructing a precise pharmaceutical service system for heart transplant patients, can improve the safety and effectiveness of medication for heart transplant patients, and has important clinical value.

ELIGIBILITY:
Inclusion Criteria:

* Patients after heart transplantation

Exclusion Criteria:

* Graft failure or death after surgery
* Patients who have received two or more organ transplants
* Patients with incomplete clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing allogeneic orthotopic heart transplantation under cardiopulmonary bypass (CPB) for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Steady state whole blood trough concentration of tacrolimus | Three days after the first dose or adjustment, blood samples were taken 2 hours before the next dose to measure the steady state whole blood trough concentration of tacrolimus(From admission to discharge, assessed up to 2 months)
  Steady state whole blood trough concentration is a commonly used therapeutic drug monitoring indicator for tacrolimus.

CONTACTS AND LOCATIONS:
Overall Officials: Junrong Zhu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Pharmacy Department of Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No